CLINICAL TRIAL: NCT01568593
Title: Comparison of the Efficacy and Safety of T2750 and Vismed® in the Treatment of Moderate to Severe Dry Eye Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Laboratoires Thea (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LT2750-PIII-10/11
Record Dates: First submitted 2012-03-29; First posted 2012-04-02 (Estimated); Results first posted 2014-10-27 (Estimated); Last update posted 2016-04-04 (Estimated); Status verified 2014-10

CONDITIONS: Dry Eye Syndromes
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- T2750 (Experimental)
  Interventions: Device: T2750
- Vismed (Active Comparator)
  Interventions: Device: Vismed

INTERVENTIONS:
Device: T2750 — 1 drop in each eye 3 to 6 times daily during 84 days
  Arms: T2750
Device: Vismed — 1 drop in each eye 3 to 6 times daily during 84 days
  Arms: Vismed

SUMMARY:
Comparison of the efficacy and safety of T2750 and Vismed® in the treatment of moderate to severe Dry Eye Syndrome

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent
* Male or female aged from ≥ 18 years old.
* Known Dry Eye Syndrome requiring artificial tears within the last 3 months prior to study selection.

Exclusion Criteria:

* Best far corrected visual acuity < 1/10
* Severe blepharitis
* Severe Dry Eye
* Eyelid malposition
* Known hypersensitivity to one of the components of the study medications or test products.
* Pregnant or breast-feeding woman.
* Woman of childbearing age (neither menopausal, nor hysterectomised, nor sterilized) not using effective contraception (oral contraceptives, intra-uterine device, contraceptive implant or condoms).
* Inability of patient to understand the study procedures and thus inability to give informed consent.
* Non compliant patient (e.g. not willing to attend the follow-up visits, way of life interfering with compliance).
* Already included once in this study.
* Patient under guardianship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2012-03; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Paris, France

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | T2750 | Vismed
Started | 48 | 45
Completed | 41 | 42
Not Completed | 7 | 3
Not completed — Lack of Efficacy | 4 | 1
Not completed — Adverse Event | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | T2750 | Vismed | Total
Number analyzed (Participants) | 48 | 45 | 93
Age, Continuous [Mean (Standard Deviation); unit: years] | 62 (11.2) | 63.6 (10) | 62.8 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 38 | 78
  Male | 8 | 7 | 15
Time from the dry eye diagnosis [Mean (Standard Deviation); unit: years] | 7.18 (6.98) | 6.2 (5.41) | 6.71 (6.25)

OUTCOME MEASURES:

1. Primary Outcome: Global Ocular Staining (With Oxford Scale - Ranges :0-15)
Description: Change from baseline in the worse eye on Day 35 (decrease of Oxford score = better outcome)
Time Frame: Baseline and 35 days
Population: Per Protocol Population
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | T2750 | Vismed
Number analyzed (Participants) | 42 | 40
scores on a scale | -1.8 (2.2) | -2 (1.4)

ADVERSE EVENTS:
Arm/Group | T2750 | Vismed
Serious Adverse Events (participants affected / at risk) | 1/48 | 0/45
Other Adverse Events (participants affected / at risk) | 0/48 | 0/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | T2750 (N=48) | Vismed (N=45)
Depression (Psychiatric disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All the results of the Trial are the sole and exclusive property of THEA, and cannot be used in whatever from without prior written agreement of THEA